CLINICAL TRIAL: NCT03652077
Title: A Phase 1, Open-Label, Dose-Escalation, Safety and Tolerability Study of INCAGN02390 in Participants With Select Advanced Malignancies
Brief Title: A Safety and Tolerability Study of INCAGN02390 in Select Advanced Malignancies
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Incyte Corporation (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: INCAGN 2390-101
Record Dates: First submitted 2018-08-28; First posted 2018-08-29 (Actual); Last update posted 2021-11-15 (Actual); Status verified 2021-11

CONDITIONS: Cervical Cancer; Gastric Cancer; Stomach Cancer; Gastroesophageal Junction Cancer; Esophageal Cancer; Hepatocellular Carcinoma; Melanoma; Uveal Melanoma; Merkel Cell Carcinoma; Mesothelioma; MSI; Non-small Cell Lung Cancer; NSCLC; Ovarian Cancer; Squamous Cell Carcinoma of the Head and Neck; Small Cell Lung Cancer; Renal Cell Carcinoma; RCC; Triple-negative Breast Cancer; Urothelial Carcinoma; Mismatch Repair Deficiency
Keywords: Advanced malignancies; immunoglobulin (Ig)G1k monoclonal antibody; T-cell immunoglobulin and mucin domain 3 (TIM-3)
MeSH Terms: conditions — Uterine Cervical Neoplasms; Stomach Neoplasms; Esophageal Neoplasms; Carcinoma, Hepatocellular; Melanoma; Uveal Melanoma; Carcinoma, Merkel Cell; Mesothelioma; Carcinoma, Non-Small-Cell Lung; Ovarian Neoplasms; Squamous Cell Carcinoma of Head and Neck; Small Cell Lung Carcinoma; Carcinoma, Renal Cell; Triple Negative Breast Neoplasms; Carcinoma, Transitional Cell; Turcot syndrome

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- INCAGN02390 (Experimental)
  Interventions: Drug: INCAGN02390

INTERVENTIONS:
Drug: INCAGN02390 — Part 1: INCAGN02390 at the protocol-defined starting dose administered every 2 weeks (Q2W), with dose escalation in 7 total cohorts to determine the maximum tolerated dose or PAD.

SUMMARY:
The purpose of this study is to determine the safety, tolerability, and preliminary efficacy of INCAGN02390 in participants with select advanced malignancies.

ELIGIBILITY:
Inclusion Criteria:

* Participants with locally advanced or metastatic tumors who are not eligible for any available therapy likely to convey clinical benefit (locally advanced disease must not be amenable to resection with curative intent).
* Participants who have disease progression after treatment with available therapies that are known to confer clinical benefit or who are intolerant to treatment.
* Willingness and ability to safely undergo pretreatment and on-treatment tumor biopsies (core or excisional).
* Eastern Cooperative Oncology Group performance status 0 or 1.
* Willingness to avoid pregnancy or fathering children based on protocol-defined criteria.

Exclusion Criteria:

* Laboratory values at screening outside the protocol-defined ranges.
* Administration of colony-stimulating factors within 14 days before Study Day 1.
* Receipt of anticancer medications or investigational drugs within protocol-defined intervals before the first administration of study drug.
* Receipt of a live vaccine within 30 days of planned start of study drug.

Note: Examples of live vaccines include, but are not limited to, the following: measles, mumps, rubella, chicken pox/zoster, yellow fever, rabies, Bacillus Calmette-Guérin, and typhoid vaccine. Seasonal influenza vaccines for injection are generally killed virus vaccines and are allowed; however, intranasal influenza vaccines are live-attenuated vaccines and are not allowed.

* Active autoimmune disease that required systemic treatment in the past (ie, with use of disease-modifying agents, corticosteroids, or immunosuppressive drugs).
* Known active central nervous system metastases and/or carcinomatous meningitis.
* Known additional malignancy that is progressing or requires active treatment, or history of other malignancy within 2 years of study entry with the exception of cured basal cell or squamous cell carcinoma of the skin, superficial bladder cancer, prostate intraepithelial neoplasm, carcinoma in situ of the cervix, or other noninvasive or indolent malignancy, or cancers from which the participant has been disease-free for > 1 year, after treatment with curative intent.
* Evidence of active, noninfectious pneumonitis or history of interstitial lung disease.
* Active infection requiring systemic therapy.
* Evidence of active HBV or HCV infection.
* Known history of HIV (HIV 1/2 antibodies).
* Known allergy or reaction to any component of study drug or formulation components.
* Prior treatment with an anti-TIM-3 antibody for any indication.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2018-09-24 (Actual); Primary Completion 2021-08-18 (Actual); Study Completion 2021-08-18 (Actual)

PRIMARY OUTCOMES:
Number of treatment-emergent adverse events | Up to 12 months
  Adverse events reported for the first time or worsening of a pre-existing event after first dose of study drug.
Maximum tolerated dose or pharmacologically active dose (PAD) of INCAGN02390 (Part 1 only) | Up to approximately 1 month
  PAD defined as a dose that achieves a level of receptor occupancy considered to be biologically active.

SECONDARY OUTCOMES:
Cmax of INCAGN02390 | Up to 12 months
  Maximum observed plasma or serum concentration.
Tmax of INCAGN02390 | Up to 12 months
  Time to maximum concentration.
Cmin of INCAGN02390 | Up to 12 months
  Minimum observed plasma or serum concentration over the dose interval.
AUC0-t of INCAGN02390 | Up to 12 months
  Area under the plasma or serum concentration-time curve from time = 0 to the last measurable concentration at time = t.
Objective response rate | Up to 12 months
  Defined as the percentage of participants having complete response (CR) or partial response (PR) determined by investigator assessment of radiographic disease per Response Evaluation Criteria in Solid Tumors (RECIST) v1.1.
Duration of response | Up to 12 months
  Defined as time from earliest date of disease response (CR or PR) until earliest date of disease progression (determined by investigator assessment of radiographic disease per RECIST v1.1) or death from any cause, if occurring sooner than progression.
Disease control rate | Up to 12 months
  Defined as percentage of participants having CR, PR, or stable disease as best on-study response.
Progression-free survival | Up to 12 months
  Defined as the time from date of first dose of study drug until the earliest date of disease progression (determined by investigator assessment of objective radiographic disease per RECIST v1.1) or death from any cause if occurring sooner than progression.
Level of binding of INCAGN02390 to TIM-3 | Up to approximately 3 months
  Assessed from participant whole blood samples.
Immunogenicity of INCAGN02390 | Up to 12 months
  Defined as the occurrence of specific ADA to INCAGN02390.

CONTACTS AND LOCATIONS:
Overall Officials: Nawel Bourayou, MD, Study Director — Incyte Corporation
Locations (4):
- United States (4):
  - The Angeles Clinical and Research Institute, Los Angeles, California
  - University of Mississippi, Jackson, Mississippi
  - Hackensack Medical Center, Hackensack, New Jersey
  - Carolina BioOncology, Huntsville, North Carolina

IPD SHARING:
Plan to Share IPD: No